

### Statistical Analysis Plan

NCT Number: NCT05107960

Title: Special Drug Use Surveillance; AZILVA Tablets and AZILVA Granules 1% in

Pediatric Use

Study Number: TAK-536-4001

Document Version and Date: Original version / 23-OCT-2024

Certain information within this document has been redacted (ie, specific content is masked irreversibly from view) to protect either personally identifiable information or company confidential information.

Note; This document was translated into English as the language on original version was Japanese.

# intercial use only and subject to the applicable Terms of Use applicable only and subject to the applicable only applicable only and subject to the applicable only applica Statistical Analysis Plan

Product Name

Surveillance Title

**Sponsor** 

Head of Biostatistics Office,

Property of Lakeda. For non' Takeda Pharmaceutical Company Limited

Ver. 1: Prepared on October 23, 2024

### Table of Contents

| 1 | Definitions of Terms | | | |
|---|---|---|---|---|
| | 1.1 | Lis | t of Terms and Abbreviations | 3 |
| | 1.2 | Ana | alysis Sets | 6 |
| | 1.3 | Nu | mber of Digits Displayed | 7 |
| | 1.4 | Saf | ety Specification | 8 |
| 2 | | | | |
| | 2.1 | .1 Disposition of Cases | | |
| 3 | Pati | ient ( | Characteristics | .10 |
| | 3.1 Patient Characteristics | | | |
| 4 | 2.1 Disposition of Cases Patient Characteristics 3.1 Patient Characteristics Comorbidities | | | |
| | 4.1 | Lis | t of Comorbidities | . 11 |
| 5 | Treatment | | | |
| | 5.1 | | | |
| | | Medication Other Than Antihypertensives) Treatment Status | | |
| 6 | Saf | etv I | nformation | .12 |
| | 6.1 | Inc | idence of Adverse Events and Adverse Reactions/Infections | .12 |
| | | .1.1 | Incidence of Adverse Events | .12 |
| | 6. | .1.2 | | .14 |
| | 6.2 Incidence of Adverse Events and Adverse Reactions/Infections Corresponding to Safety | | | |
| | | | pecification | .15 |
| | 6. | .2.1 | | |
| | 6. | .2.2 | 76 | |
| | 6.3 | Inc | idence of Adverse Events and Adverse Reactions/Infections in Patients Excluded | |
| | | Fr | rom Safety Analysis | .16 |
| | 6. | .3.1 | Incidence of Adverse Events in Patients Excluded From Safety Analysis | .16 |
| | 6. | .3.2 | Incidence of Adverse Reactions/Infections in Patients Excluded from Safety | |
| | | 7 | Analysis | .16 |
| | 6.4 | | idence of Adverse Reactions/Infections Leading to Discontinuation of Azilsartan | |
| , | <0. | • | reatment | .16 |
| <i>y</i> | 6. | .4.1 | Incidence of Adverse Reactions/Infections Leading to Discontinuation of Azilsartan | |
| | | | Treatment | .16 |
| | 6.5 | Inc | idence of Adverse Events and Adverse Reactions/Infections by Seriousness, Time of | |
| | | | nset, Outcome, and Causal Relationship to Azilsartan | .17 |
| | 6. | .5.1 | Incidence of Adverse Events by Seriousness, Time of Onset, Outcome, and Causal | |
| | | | Relationship to Azilsartan | 17 |

### 1 Definitions of Terms

### 1.1 List of Terms and Abbreviations

- Azilsartan: Azilsartan is the generic term for Azilva Tablets and Azilva Granules 1%.
- Adverse event: An adverse event occurring after the administration of azilsartan.
- Adverse reactions, etc.: An abbreviation for the term "adverse reactions/infections." Adverse
  events other than any assessed as "not related" to azilsartan by investigators. In this statistical
  analysis plan, "adverse reactions/infections" will be used in the titles, and "adverse reactions,
  etc." will be used in the text and tables.
- Serious adverse event: An adverse event assessed as being "serious" by investigators Based on
  the Important Medical Events List, events listed in the MedDRA Code List (PT code) will be
  handled as serious even if assessed by investigators as "non-serious."
- "Related" to azilsartan: An adverse event with a causal relationship other than "unrelated" to azilsartan.
- "Not related" to azilsartan: An adverse event for which a causal relationship to azilsartan was ruled out.
- Summary statistics: A collective term for sample size, mean, standard deviation, maximum, minimum, and quartile values.
- Patients for whom no CRFs were collected: Enrolled patients for whom no CRFs were collected.
- Patients for whom CRFs were collected: Enrolled patients for whom CRFs were collected.
- Age: Age (at the time azilsartan is prescribed) will be used. If age (at the time azilsartan is
  prescribed) is missing, age will be derived as follows.

If the birth month is prior to the month at the start of azilsartan treatment, age will be calculated as the year at the start of azilsartan treatment - birth year - 1. If the birth month is the same as or after the month at the start of azilsartan treatment, age will be calculated as the year at the start of azilsartan treatment - birth year. However, if the birth month is unknown, it will be calculated as January.

• Duration of azilsartan treatment (days): End of azilsartan treatment date - start of azilsartan treatment date + 1

Wash out periods, if any, will be excluded from the duration of azilsartan treatment (days).

If the end of azilsartan treatment date is unknown or treatment continues past the end of the observation period, the vital signs/body weight measurement date or the laboratory tests date, whichever is last, will be used as the end of azilsartan treatment date.

Antihypertensives \*Within 3 months prior to start of treatment:

Antihypertensives taken prior to start of azilsartan treatment (that are used with or without azilsartan). Any antihypertensive meeting any of the following conditions that is reported in the "Concomitant medication (antihypertensive other than azilsartan) treatment status" section of the CRF. The CRF states the following: "Document any antihypertensives other than azilsartan that are used from 3 months before the start of azilsartan treatment up to 12 months after the start of azilsartan treatment or until discontinued. Any antihypertensives that are discontinued within 3 months before the start of azilsartan treatment should also be documented." Therefore, no statistical analysis of the 3-month period prior to azilsartan treatment will be performed in the analysis.

- · Start of treatment date before start of azilsartan treatment date
- · End of treatment date before start of azilsartan treatment date
- Ongoing since 3 months before the start of azilsartan treatment
- Concomitant medication (antihypertensive other than azilsartan) \*After the start of azilsartan treatment:

Antihypertensives administered during azilsartan treatment period. Any antihypertensive meeting any of the following conditions that is reported in the "Concomitant medication (antihypertensive other than azilsartan) treatment status" section of the CRF.

- Start of treatment date is on or after start of azilsartan treatment date, or end of treatment date is on or after start of azilsartan treatment date
- Start of treatment date is prior to start of azilsartan treatment date, and continues past end of observation period
- Ongoing since 3 months before start of azilsartan treatment, and continues past end of observation period
- Time of onset of adverse event (or adverse reaction, etc.): Calculated as the date of onset of adverse event (or adverse reaction, etc.) start of azilsartan treatment date + 1.
- Duration of disease:

Actual number (unit: year) = (year when first azilsartan dose initiated - year when hypertension was diagnosed) + (month when the first azilsartan dose initiated - month when hypertension was diagnosed)/12 (rounded off to first decimal place).

If the month of diagnosis is unknown, it will be calculated as January of the reported year. If the year of diagnosis is unknown, it will be considered to be missing data.

• BMI (kg/m<sup>2</sup>): Calculated as body weight (kg)/height (m)<sup>2</sup> (rounded off to first decimal place).

Property of Takeda: For non-commercial use only and subject to the applicable Terms of tuse • eGFR (mL/min/1.73m<sup>2</sup>): Calculated using the following formula for estimating GFR in Japanese children, as reported by the Pediatric Chronic Kidney Disease Task Force. The most recently

5

### 1.2 **Analysis Sets**

In this surveillance, the "safety analysis set" and the "efficacy analysis set" will be used as the analysis sets. These are defined as follows.

### • Safety analysis set

the applicable rerms of Use This is defined as "patients for whom the CRF is locked, who receive at least one dose of azilsartan and can be assessed for safety." Patients for whom the CRF is locked will be excluded from the safety analysis set if the following conditions are applicable.

- No azilsartan treatment
- Enrolled 15 or more days after date on which azilsartan is first prescribed
- Adverse event status unknown

### • Efficacy analysis set

Property of Takeda. For non-commercial use only and subtraction of takeda. This is defined as "patients of the safety analysis set who have no major protocol violations and can be assessed for efficacy." Patients of the safety analysis set will be excluded from the efficacy

### **Number of Digits Displayed**

### Percentages (%)

Incidence of adverse events or adverse reactions, etc.:

All others:

### Summary statistics

Mean, 1st quartile, median, 3rd quartile:

Standard deviation:

ean, 1st quartile, median, 3rd quartile:
Round off the second digit of the source data and display to the first digit of the source data and display to the second digit of the source data and display to the second digit of the nimum, maximum:

Display the same number of digits as the Minimum, maximum:

### Confidence interval

ended of Takeda. For non-commercial use only and subject to Round off the third digit of the source data and display to the second digit of the source data.

7

### 1.4 Safety Specification

- Important identified risks
- Hypotension-related events: Events corresponding to MedDRA PT codes 10005731 (blood pressure ambulatory decreased), 10005737 (blood pressure diastolic decreased), 10066077 (diastolic hypotension), 10053356 (blood pressure orthostatic decreased), 10005734 (blood pressure decreased), 10005758 (blood pressure systolic decreased), 10084013 (post procedural hypotension), 10062300 (procedural hypotension), 10013573 (dizziness), 10013578 (dizziness postural), 10021097 (hypotension), 10031127 (orthostatic hypotension), 10036653 (presyncope), 10042772 (syncope), 10047340 (vertigo), 10047348 10013578 (dizziness postural), 10021097 (hypotension), 10031127 (orthostatic property of Takeda. For non-commercial use only and subject to (vertigo positional), 10024855 (loss of consciousness), 10012373 (depressed level of consciousness), 10009192 (circulatory collapse), 10040560 (shock), 10040581 (shock

### Number of Surveillance Site, Number of Enrolled Patients, and Patient Disposition

### 2.1 **Disposition of Cases**

All enrolled patients (enrolled patients) Analysis population:

Analytical parameters: Enrolled patients

Surveillance sites

Patients for whom no CRFs

were collected

Patients for whom CRFs

were collected

Patients excluded from

safety analysis\*

[No azilsartan treatment, enrolled 15 or more Reason for exclusion (counted more than once)

days after date on which azilsartan is first

prescribed; adverse event status unknown]

Safety analysis set

Patients excluded from

efficacy analysis\*

[Inclusion criteria violation [discovered after Reason for exclusion

(counted more than once) the fact],

Exclusion criteria violation [discovered

after the fact]]

Efficacy Analysis Set

Analysis methods:

The following analyses will be performed for the above analytical parameters, and a patient disposition chart will be prepared.

The number of surveillance sites will also be shown for enrolled patients.

The same site having different clinical departments in the surveillance will be counted as one site.

If there are no reasons for excluding any patients, 0 subjects will be displayed.

Listings will be prepared in which the number of patients excluded from the safety and efficacy analyses will be tabulated by each reason for exclusion.

Property of Takeda. For nor, \*"Patients excluded from safety analysis" refers to patients for whom CRFs are collected who are excluded from the "safety analysis set." Similarly, "patients excluded from efficacy analysis" refers to patients in the "safety analysis set" who are excluded from the "efficacy analysis set."

> (1) Frequency tabulations

### 3 **Patient Characteristics**

### **Patient Characteristics** 3.1

Analysis population: Safety analysis set

Sex Analytical parameters:

Age (years)

Body weight (kg)

[Min <= - <20.0, 20.0 <= - <30.0, 30.0] <= - <40.0, 40.0 <= - <50.0, 50.0 <= - <60.0, 60.0 <= - <70.0, 70.0 <= < 80.0, 80.0 <= - <= Max] [Min <= - <15.0, 15.0 <= - <18.0, 18.0] <= - <21.0, 21.0 <= - <24.0, 24.0 <= - <27.0, 27.0 <= - <= Max]Outpatient, inpatient BMI  $(kg/m^2)$ 

Inpatient/outpatient status

baseline)

Comorbidities

[No, yes, unknown] Medical history

Predisposition to hypersensitivity [No, yes, unknown]

[Min <= - <30, 30 <= - <45, 45 <= - <60, eGFR (mL/min/1.73m<sup>2</sup>)

 $60 \le - \le 90, 90 \le - \le Max$ 

Systolic blood pressure (mmHg)

Diastolic blood pressure (mmHg)

Pulse rate (bpm)

Disease duration (years) [Min <= - <1, 1 <=- <2, 2 <= - <3, 3 <=

-<4, 4<=-<=Max

Antihypertensive treatment

\*Within 3 months prior to start of [No, yes]

treatment

Analysis methods: Frequency tabulations of discrete data will be prepared and summary

statistics of categorical data will be calculated for the above analytical

parameters.

### **Comorbidities**

### **List of Comorbidities** 4.1

Analysis population: Safety analysis set

Analytical parameters: Case number

Disease name

Analysis methods: Listings of the above analytical parameters will be prepared.

### **Treatment**

### arta applica Azilsartan and Concomitant Medication (Antihypertensives Other Than Azilsartan, and 5.1 **Medication Other Than Antihypertensives) Treatment Status**

Analysis population: Safety analysis set

Analytical parameters: Case number

Initial azilsartan dose (mg)

Change in daily dose

Mean azilsartan daily dose (mg)

Duration of azilsartan treatment (days)

Discontinuation of azilsartan

Reason for discontinuation of azilsartan

Concomitant medication (antihypertensive other than azilsartan) treatment

Breakdown of concomitant medication (antihypertensive other than

Concomitant medication (other than antihypertensive) treatment

Breakdown of concomitant medication (other than antihypertensives)

### **Safety Information**

If 0 adverse events are reported in the safety analysis set, no tabulations will be prepared for Sections 6.1.2, 6.2, 6.4, 6.5, and 6.6. If 0 patients are excluded from safety analysis, no tabulations will be prepared for Section 6.3. If 1 or more patients are excluded from safety analysis and 0 adverse Adverse events

The following analyses will be performed for the above analytical parameter.

(1) Number of patients with adverse events

2) Number of adverse events

3) Incidence of events are reported, tabulations will be prepared for Section 6.3.1, and no tabulations will be prepared for Section 6.3.2.

### 6.1 **Incidence of Adverse Events and Adverse Reactions/Infections**

### 6.1.1 **Incidence of Adverse Events**

Analysis population: Analytical parameters:

cx to the appl Analysis methods:

(4) Type of adverse events

Each analysis will be carried out as follows

[Number of patients with adverse events]

The number of patients who experience adverse events.

[Number of adverse events]

The number of adverse events that occur. If the same adverse event occurs more than once in the same patient, the total number of events will be tabulated.

This will be calculated as the number of patients with adverse events divided by the number of patient. divided by the number of patients in the safety analysis set multiplied by 100.

### [Type of adverse events]

- Property of Takeda. For non-Adverse events will be coded using the MedDRA/J. These will be broadly classified by SOC, and will be tabulated by PT within those classifications. Those in the SOC of "investigations" will be tabulated by HLGT (sorted in ascending order of HLGT code, but without listing the codes) and tabulated by PT.
  - In SOC tabulations, the number of patients with adverse events and the incidence of adverse events will be documented in order of SOC international consensus. If the same SOC occurs more than once in the same patient, the patient will be counted only once for that SOC.

In PT tabulations, the number of patients with adverse events and the incidence of adverse events will be documented in ascending order of

Property of Takeda: For non-commercial use only and subject to the applicable Terms of tuse

### 6.1.2 Incidence of Adverse Reactions/Infections

Analysis population: Safety analysis set

Analytical parameters: Adverse reactions, etc.

Analysis methods: The following analyses will be performed for the above analytical

parameter.

(1) Number of patients with adverse reactions, etc.

- (2) Number of adverse reactions, etc.
- (3) Incidence of adverse reactions, etc.
- (4) Types of adverse reactions, etc.

Each analysis will be carried out as follows.

[Number of patients with adverse reactions, etc.]

· The number of patients who experience adverse reactions, etc.

[Number of adverse reactions, etc.]

The number of adverse reactions, etc. that occur. If the same adverse reaction, etc. occurs more than once in the same patient, the total number of events will be tabulated.

[Incidence of adverse reactions, etc.]

This will be calculated as the number of patients with adverse reaction, etc. divided by the number of patients in the safety analysis set multiplied by 100.

[Types of adverse reactions, etc.]

Adverse reactions, etc. will be coded using the MedDRA/J. These will be broadly classified by SOC, and will be tabulated by PT within those classifications. Those in the SOC of "investigations" will be tabulated by HLGT (sorted in ascending order of HLGT code, but without listing the codes) and tabulated by PT.

- In SOC tabulations, the number of patients with adverse reactions, etc. and the incidence of adverse reactions, etc. will be documented in order of SOC international consensus. If the same SOC occurs more than once in the same patient, the patient will be counted only once for that SOC.
- · In PT tabulations, the number of patients with adverse reactions, etc. and the incidence of adverse reactions, etc. will be documented in ascending order of PT code. If the same PT occurs more than once in the same patient, the patient will be counted only once for that PT.

### **6.2** Incidence of Adverse Events and Adverse Reactions/Infections Corresponding to Safety Specification

### 6.2.1 Incidence of Adverse Events Corresponding to Safety Specification

Analysis population: Safety analysis set

Analytical parameters: Adverse events corresponding to the safety specification (important

identified risks)

Stratification factors: Seriousness [Serious, non-serious]

Analysis methods: Stratified analysis of the above, by stratification factor and by risk, will be

performed in the same manner as in Section 6.1.1. If the same SOC/PT occurs more than once in the same patient, the patient will be counted only

once for that SOC/PT. However, if the seriousness of the events is different,

the events will each be counted as serious or non-serious event, respectively. In addition, the risk will be assessed per the definitions

specified in 1.4 Safety Specification.

### 6.2.2 Incidence of Adverse Reactions/Infections Corresponding to Safety Specification

Analysis population: Safety analysis set

Analytical parameters: Adverse reactions, etc. corresponding to the safety specification (important

identified risks)

Stratification factors: Seriousness [Serious, non-serious]

Analysis methods: Stratified analysis of the above, by stratification factor and by risk, will be

performed in the same manner as in Section 6.1.2. If the same SOC/PT occurs more than once in the same patient, the patient will be counted only once for that SOC/PT. However, if the seriousness of the events is different,

the events will each be counted as serious or non-serious event,

respectively. In addition, the risk will be assessed per the definitions

specified in 1.4 Safety Specification.

### 6.3 Incidence of Adverse Events and Adverse Reactions/Infections in Patients Excluded From Safety Analysis

### 6.3.1 Incidence of Adverse Events in Patients Excluded From Safety Analysis

Analysis population:

Analytical parameters:

Analysis methods:

### Incidence of Adverse Reactions/Infections in Patients Excluded from Safety Analysis population: Patients excluded from safety analysis al parameters: Adverse reactions, etc. methods: The above will! 6.3.2

Analysis population:

Analytical parameters:

Analysis methods:

### Incidence of Adverse Reactions/Infections Leading to Discontinuation of Azilsartan 6.4 **Treatment**

### Incidence of Adverse Reactions/Infections Leading to Discontinuation of Azilsartan 6.4.1 **Treatment**

Safety analysis set Analysis population:

Adverse reactions, etc. leading to discontinuation of azilsartan treatment Analytical parameters:

The above will be analyzed in the same manner as in Section 6.1.2.

### 6.5 Incidence of Adverse Events and Adverse Reactions/Infections by Seriousness, Time of Onset, Outcome, and Causal Relationship to Azilsartan

### 6.5.1 Incidence of Adverse Events by Seriousness, Time of Onset, Outcome, and Causal Relationship to Azilsartan

Analysis population: Safety analysis set Analytical parameters: Adverse events

Stratification factors: Total

> [Serious, non-serious] Seriousness

Time of onset (day)

[1 <= - <= 14, 15 <= - <= 28, 29 <= - <= 42, 43 <= - <= 56, 57 <= <= 70, 71 <= - <= 84, 85 <= - <= Max]

[1 <= - <= 84, 85 <= = 168, 169 <= -<= 252, 253 <= - <= 336, 337 <= - <= 420, 421 <= - <= Max]

Outcome [Resolved, Resolving, Not resolved,

Resolved with sequelae, Death (due to

this event), Unknown]

Causal relationship to [Related, unrelated]

azilsartan

Stratified analysis of the above by stratification factor will be performed in Analysis methods:

the same manner as in Section 6.1.1. If the same SOC/PT occurs more than

once in the same patient, the patient will be counted only once for that

SOC/PT. However, SOCs that are the same will be handled as one in the

following order of priority, and PTs that are the same will be handled as

one per the details of one of the stratification factors in the following order

of priority.

Seriousness: Serious → Non-serious

Time of onset 1 (days): 1-14 days  $\rightarrow$  15-28 days  $\rightarrow$  29-42 days  $\rightarrow$  43-56

 $days \rightarrow 57-70 \ days \rightarrow 71-84 \ days \rightarrow \ge 85 \ days$ 

Time of onset 2 (days): 1-84 days  $\rightarrow$  85-168 days  $\rightarrow$  169-252 days  $\rightarrow$  253-

336 days  $\rightarrow$  337-420 days  $\rightarrow$   $\geq$  421 days

Outcome: Death (due to this event)  $\rightarrow$  Resolved with sequelae  $\rightarrow$  Not

 $resolved \rightarrow Resolving \rightarrow Resolved \rightarrow Unknown$ 

Causal relationship to azilsartan: Related → Not related

### 6.5.2 Incidence of Adverse Reactions/Infections by Seriousness, Time of Onset, and

### Outcome

Safety analysis set Analysis population: Analytical parameters: Adverse reactions, etc.

Stratification factors: Total

> Seriousness [Serious, non-serious]

Time of onset (day)

[1 <= - <= 14, 15 <= - <= 28, 29 <= - <= 42, 43 <= - <= 56, 57 <= - <= 70, 71 <= - <= 84, 85 <= - <= Max]

[1 <= - <= 84, 85 <= - <= 168, 169 <= -

<= 252, 253 <= - <= 336, 337 <= - <=

420, 421 <= - <= Max]

[Resolved, Resolving, Not resolved, Outcome

Resolved with sequelae, Death (due to

this event), Unknown]

Stratified analysis of the above by stratification factor will be performed in Analysis methods:

the same manner as in Section 6.12. If the same SOC/PT occurs more than

once in the same patient, the patient will be counted only once for that

SOC/PT. However, SOCs that are the same will be handled as one in the

following order of priority, and PTs that are the same will be handled as

one per the details of one of the stratification factors in the following order

of priority.

Seriousness: Serious → Non-serious

Time of onset 1 (days): 1-14 days  $\rightarrow$  15-28 days  $\rightarrow$  29-42 days  $\rightarrow$  43-56

 $days \rightarrow 57-70 days \rightarrow 71-84 days \rightarrow \ge 85 days$ 

Time of onset 2 (days): 1-84 days  $\rightarrow$  85-168 days  $\rightarrow$  169-252 days  $\rightarrow$  253-

336 days  $\rightarrow$  337-420 days  $\rightarrow$   $\geq$  421 days

Outcome: Death (due to this event)  $\rightarrow$  Resolved with sequelae  $\rightarrow$  Not

 $resolved \rightarrow Resolving \rightarrow Resolved \rightarrow Unknown$ 

### 6.6 Incidence of Adverse Reactions/Infections by Patient Characteristics and Treatment **Factors**

## , yes] to the applicable Terms of Use 6.6.1 List of Adverse Reactions/Infections by Patient Characteristics and Treatment

### **Factors**

Analysis population: Safety analysis set

Analytical parameters: Case number

Sex

Age (years)

Comorbidities

Breakdown of comorbidities Initial azilsartan dose (mg) Antihypertensive treatment

\*Within 3 months prior to start of

treatment

Date of onset

SOC PT

Hypotension-related events

Seriousness [Serious, non-serious]

Outcome [Resolved, Resolving, Not resolved,

Resolved with sequelae, Death (due

to this event), Unknown]

discontinuation

[Yes, no]

azilsartan treatment

of Takeda. For none Listings of the above analytical parameters will be prepared for patients

experiencing adverse reactions, etc.

19

### 7 Efficacy Information

### 7.1 Changes in Blood Pressure Over Time

Analysis population: Efficacy analysis set

Analytical parameters: Systolic blood pressure (mmHg), diastolic blood pressure (mmHg)

Analysis methods: For each of the above analytical parameters, summary statistics will be

calculated for laboratory values at each assessment time point (baseline and

after 1 month of azilsartan treatment to after 12 months of azilsartan

treatment) as well as changes (laboratory values at each assessment time point after baseline-laboratory values at baseline). Listings will be shown rather than summary statistics when the efficacy analysis set includes 2 or

fewer patients. Changes over time in laboratory values will also be plotted

individually.

### 7.2 List of Factors Potentially Affecting Efficacy

Analysis population: Efficacy analysis set

Analytical parameters: Case number

Sex [Male, female]

Age (years)

Comorbidities [No, yes]

Breakdown of comorbidities Initial azilsartan dose (mg) Antihypertensive treatment

\*Within 3 months prior to start of [No, yes]

treatment

Breakdown of antihypertensive

treatment \*Within 3 months prior

to start of treatment

Assessment time point

Systolic blood pressure (mmHg)

Diastolic blood pressure (mmHg)

Analysis methods: Listings of the above analytical parameters will be prepared.

### Incidence of Adverse Reactions/Infections in Supplementary Pharmacovigilance Plan

### 8.1 Incidence of Adverse Reactions/Infections in Supplementary Pharmacovigilance Plan (Attachment Form 12)

Analysis population: Safety analysis set

Lerins of Use Analytical parameters: Adverse reactions, etc. corresponding to the safety specification (important

identified risks)

Stratification factors: Seriousness [Serious, non-serious]

Analysis methods: The above analytical parameters will be analyzed, stratified by

> stratification factor, according to (Notes) 1 through 4 of Attachment Form 12 in PSEHB/PED Reexamination Notification No. 0325-10, dated March

25, 2020.

Number of patients and incidence (1)

Property of Takeda. For non-commercial use only and subject of Takeda. The risk terms that are used and the order in which they are listed will be based on the definitions given in the Important Identified Risks section.

### Incidence of Adverse Reactions/Infections in Post-Marketing Surveillance

### Incidence of Adverse Reactions/Infections in Post-Marketing Surveillance (Attachment 9.1 **Form 15)**

Analysis population: Safety analysis set Analytical parameters: Adverse reactions, etc.

The following analyses will be performed for the above analytical Analysis methods: parameter.

- (1) Status of post-marketing surveillance
  - 1) Number of patients in safety analysis set
  - 2) Number of patients with adverse reactions, etc.
  - Incidence of adverse reactions, etc.
- Types of adverse reactions, etc. (2)
  - Number of patients with adverse reactions, etc. and incidence (by SOC)
  - Number of patients with adverse reactions, etc. and incidence 2) (by PT)

Each analysis will be carried out as follows.

[Number of patients with adverse reactions, etc.]

The number of patients who experience adverse reactions, etc.

[Incidence of adverse reactions, etc.]

This will be calculated as the number of patients with adverse reaction, etc. divided by the number of patients in the safety analysis set multiplied by 100.

[Types of adverse reactions, etc.]

Adverse reactions, etc. will be coded using the MedDRA/J. These will be broadly classified by SOC, and will be tabulated by PT within those classifications. Those in the SOC of "investigations" will be tabulated by HLGT (sorted in ascending order of HLGT code, but without listing the codes) and tabulated by PT.

- Property of Takedai. For non's In SOC tabulations, the number of patients with adverse reactions, etc. and the incidence of adverse reactions, etc. will be documented in order of SOC international consensus. If the same SOC occurs more than once in the same patient, the patient will be counted only once for that SOC.
  - In PT tabulations, the number of patients with adverse reactions, etc. and the incidence of adverse reactions, etc. will be documented in

Property of Takeda: For non-commercial use only and subject to the applicable Terms of tuse ascending order of PT code. If the same PT occurs more than once in the same patient, the patient will be counted only once for that PT.

### 10 Summary of Cases in Post-Marketing Surveillance

### 10.1 Summary of Cases in Post-Marketing Surveillance (File for Reexamination Data Entries)

Analysis population: Patients for whom CRFs were collected

Analytical parameters: Case number

Name of site

Sex

Age

Reason for use (disease code, disease name) Comorbidities (disease code, disease name)

Route of administration

Maximum dose

Mean dose

Units

Duration of use (duration of azilsartan treatment)

Concomitant medications (drug code, drug name)

Effect size

Adverse reactions (disease code, disease name, outcome)

CRF number

Dropped out

Reason for dropout

Analysis methods: Listings of the above analytical parameters will be prepared in accordance

> with the Guidelines for Preparation of File for Reexamination Data Entries in PSEHB/PED Reexamination Notification No. 1119-3, dated November

Property of Takedai. For non!

24

### **Document History (Version Management)**

| Version | Date | Created/Modified by | Comments |
|---------|------------|---------------------|-----------------|
| Ver. 1 | 2024.10.23 | | Ver. 1 prepared |

Property of Takeda: for non-commercial use only and subject to the applicable Terms of tuse